CLINICAL TRIAL: NCT06030336
Title: Home Health and Air Pollution Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: University of Colorado, Denver (Other); Access Sensor Technologies, LLC (Unknown)
Responsible Party: Principal Investigator, Ellison Carter, Associate Professor, Colorado State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23 - 0817
Record Dates: First submitted 2023-08-30; First posted 2023-09-11 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Indoor Air Quality

STUDY DESIGN:
Intervention Model Description: Random assignment to the intervention or control group in blocks of four households, to maintain balance in the intervention and control groups over the course of study enrollment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The Home Health Report will provide quantitative information about health-relevant pollutants (fine particulate matter, carbon dioxide, nitrogen dioxide, and volatile organic compounds), their levels compared to health-based guidelines, their potential sources, as well as no- and low-cost actions occupants could take to improve indoor air quality. The Home Health Report will be designed to maximize utility to residents. Each Home Health Report will be provided after the corresponding Home Health Box deployment. The second Home Health Box deployment will occur after the household receiving their first Home Health Report. The third and final Home Health Box deployment will occur within one month of the household receiving their second Home Health Report.
  Interventions: Behavioral: Home Health Report
- Control (No Intervention): Households in the control group will also receive three Home Health deployments spaced over several months, but will not receive Home Health Reports after the first and second deployments. At the close of their participation in the study, households in the control group will receive a comprehensive Home Health Report, including results from all three Home Health Box deployments and recommended actions occupants could take to improve their home air quality.

INTERVENTIONS:
Behavioral: Home Health Report — The Home Health Report has been described in the intervention arm description.
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to learn about whether indoor air quality will improve over time in homes where occupants receive personalized information about levels of health-relevant air pollutants that includes practical, budget-friendly, and culturally relevant recommendations on actions they can take to improve their home's air quality. The rationale for the investigators' approach is that a rigorous intervention study design will generate robust evidence on the value of the in-home environmental data. Participating homes in both the intervention and control groups will receive three, one-week Home Health Box deployments spaced six weeks apart. After each of the first two deployments, homes in the intervention group will receive a Home Health Report with personalized information about in-home levels of health-relevant air pollutants and cost-sensitive recommendations on actions occupants can take to improve their home's air quality. The investigators will (a) investigate whether and how air quality changes over time in control and intervention homes and (b) survey intervention households on the utility of the Home Health Reports.

DETAILED DESCRIPTION:
Study participation will involve: (i) an intake survey; (ii) random assignment to the intervention or control group (this will be done in blocks of 4 households, to maintain balance in the intervention and control groups over the course of study enrollment); (iii) three in-home air quality monitoring deployments with the Home Health Box; (iv) three Home Health Reports (for those randomly assigned to the intervention group) generated from data the Home Health Box provides; and (v) a follow-up survey in a subset of intervention households to investigate the value and utility of the Home Health Report. The Home Health Report will provide quantitative information about health-relevant pollutants (fine particulate matter, carbon dioxide, nitrogen dioxide, and volatile organic compounds), their levels compared to health-based guidelines, their potential sources, as well as no- and low-cost actions occupants could take to improve indoor air quality. The Home Health Report will be designed to maximize utility to residents. Each Home Health Report will be provided within approximately three to four weeks after the corresponding Home Health Box has been received from the household. The second Home Health Box deployment will occur within several weeks to one month of the household receiving their first Home Health Report. The third and final Home Health Box deployment will occur within several weeks to one month of the household receiving their second Home Health. Households in the control group will also receive three Home Health Box deployments spaced approximately four to eight weeks apart, but will not receive Home Health Reports after the first and second deployments. At the close of their participation in the study, households in both the intervention and control groups will receive a comprehensive Home Health Report, including results from all three Home Health Box deployments and recommended actions occupants could take to improve their home air quality. In total, participation in this study will last between four to six months.

ELIGIBILITY:
Inclusion Criteria:

* living in home for at least next six months

Exclusion Criteria:

* if participants will not be living in the same household within six months of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
In-Home Air Quality | from eight to up to 24 weeks
  In-home concentrations of fine particulate matter, nitrogen dioxide, and volatile organic compounds.

CONTACTS AND LOCATIONS:
Overall Officials: Ellison Carter, PhD, Principal Investigator — Colorado State University
Locations (2):
- United States (2):
  - UCHealth, Aurora, Colorado
  - Colorado State University, Fort Collins, Colorado

IPD SHARING:
Plan to Share IPD: Yes
Our human subjects work will generate a comprehensive dataset that includes information on in home exposures, in-home activities, and home air quality in the form of quantitative, reference grade information on aerosol and gas constituents in indoor air. After de-identifying these data (including location data), we will publish these data in peer-reviewed journals. We will also generate subject response data from surveys and interviews. These data will be organized, assembled, and analyzed for publication in peer-reviewed journals. Standard restrictions would apply to the secondary research use of data involving human subjects, and these data would only be made available through a written agreement with the party requesting the data, after being deidentified.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available to researchers associated with the project via the collaborating institutions as the data are being collected and for up to three years beyond the end of the study period.
Access Criteria: Researchers will be eligible for access if they are members of the overall study team.

REFERENCES:
- [Background] Tryner J, Phillips M, Quinn C, Neymark G, Wilson A, Jathar SH, Carter E, Volckens J. Design and Testing of a Low-Cost Sensor and Sampling Platform for Indoor Air Quality. Build Environ. 2021 Dec;206:108398. doi: 10.1016/j.buildenv.2021.108398. Epub 2021 Sep 28. PMID 34764540